CLINICAL TRIAL: NCT04370275
Title: Accuracy of Lung Ultrasound in the Diagnosis of covid19 Pneumonia: a Multicenter Study in the Italian Outbreak
Brief Title: Accuracy of Lung Ultrasound in the Diagnosis of covid19 Pneumonia
Acronym: POCUSars-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale di Latisana (Other)
Responsible Party: Sponsor
Other Study IDs: CEUR-2020-Os-086
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Pneumonia, Viral
Keywords: Covid-19; Lung Ultrasound; POCUS
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Is Lung Ultrasound really useful in diagnosing COVID19? What can be the usefulness of the Lung Ultrasound in the COVID19 epidemic? In the current state of the art, Sensitivity, Specificity, Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of Lung Ultrasound in the diagnosis of COVID-19 are not yet known.

Alveolar-interstitial lung diseases such as viral pneumonia and ARDS seems to have a specific ultrasound pattern that distinguishes them from bacterial pneumonia, preferentially represented by B lines, morphological irregularity of the pleural line, and small subpleural consolidations, but they could share these patterns with other pathologies, reducing specificity.

In Italy, the Lung Ultrasound represents a consolidated method for the evaluation and management of all patients who come to the ER, and what we are sure of is its high sensitivity in identifying pathological patterns.

Our preliminary data suggest that Lung Ultrasound is highly reliable not to include but to exclude the diagnosis of COVID-19 in patients with respiratory symptoms.

DETAILED DESCRIPTION:
One of the first scientific papers published on the COVID-19 epidemic in China showed that patients still asymptomatic or paucisymptomatic, positive for SARS-CoV-2 on the RT-PCR test, presented chest CT images referring to parenchymal infiltrate with a prevalent appearance at ground-glass compatible with initial COVID-19 pneumonia.

An ongoing study anticipates that the sensitivity of chest CT is higher than that of the RT-PCR molecular test for SARS-CoV-2 (performed on the pharyngeal swab or sputum) (50 out of 51, 98%, 95% CI: 90% -100% vs 36 out of 51, 71%, IC95%: 56% -83%) in the early diagnosis of COVID-19.

Recent work seems to shows that Lung Ultrasound is effective in the clinical evaluation and diagnosis of COVID-19 pneumonia.

In a previous study, in addition, sensitivity and specificity of the Lung Ultrasound in the early diagnosis of H1N1 flu pneumonia was 94.1% (32 out of 34) and 84.8% respectively (28 out of 33), with a positive predictive value of 86.5% (32 out of 37) and a negative predictive value of 93.3% (28 out of 30).

The concordance between the lung ultrasound findings and the lung lesions found on CT has recently been demonstrated ("lobe-specific" concordance equal to 87%; "lung-specific concordance" equal to 92.5 % for the right lung and 83.6% for the left lung).

These data suggest to better explore the diagnostic accuracy of the Lung Ultrasound in SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Fever and/or
* Cough and/or
* Dyspnoea

Exclusion Criteria:

* No one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People entering the Emergency Room during the SARS-CoV-2 epidemic
Sampling Method: Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-23 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value of Lung Ultrasound in the diagnosis of COVID-19 | 30 days
  Lung Ultrasound accuracy in rule-out of patients with respiratory symptoms (fever and / or cough and / or dyspnoea) during the SARS-CoV-2 epidemic compared to nasopharyngeal swab and a composite reference standards

SECONDARY OUTCOMES:
Positive Predictive Value of Lung Ultrasound in the diagnosis of COVID-19 | 30 days
  Lung Ultrasound accuracy in rule-in of patients with respiratory symptoms (fever and / or cough and / or dyspnoea) during the SARS-CoV-2 epidemic compared to nasopharyngeal swab and a composite reference standards
Sensitivity and Specificity of Lung Ultrasound in the diagnosis of COVID-19 | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Copetti, MD, Director, Principal Investigator — Ospedale di Latisana
Locations (1):
- SC Pronto Soccorso e Medicina d'Urgenza, Latisana, Udine, Italy

REFERENCES:
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Background] Tierney DM, Huelster JS, Overgaard JD, Plunkett MB, Boland LL, St Hill CA, Agboto VK, Smith CS, Mikel BF, Weise BE, Madigan KE, Doshi AP, Melamed RR. Comparative Performance of Pulmonary Ultrasound, Chest Radiograph, and CT Among Patients With Acute Respiratory Failure. Crit Care Med. 2020 Feb;48(2):151-157. doi: 10.1097/CCM.0000000000004124. PMID 31939782
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Testa A, Soldati G, Copetti R, Giannuzzi R, Portale G, Gentiloni-Silveri N. Early recognition of the 2009 pandemic influenza A (H1N1) pneumonia by chest ultrasound. Crit Care. 2012 Feb 17;16(1):R30. doi: 10.1186/cc11201. PMID 22340202
- [Background] Copetti R, Soldati G, Copetti P. Chest sonography: a useful tool to differentiate acute cardiogenic pulmonary edema from acute respiratory distress syndrome. Cardiovasc Ultrasound. 2008 Apr 29;6:16. doi: 10.1186/1476-7120-6-16. PMID 18442425
- [Background] Carley S, Dosman S, Jones SR, Harrison M. Simple nomograms to calculate sample size in diagnostic studies. Emerg Med J. 2005 Mar;22(3):180-1. doi: 10.1136/emj.2003.011148. PMID 15735264
- [Background] Tsung JW, Kessler DO, Shah VP. Prospective application of clinician-performed lung ultrasonography during the 2009 H1N1 influenza A pandemic: distinguishing viral from bacterial pneumonia. Crit Ultrasound J. 2012 Jul 10;4(1):16. doi: 10.1186/2036-7902-4-16. PMID 22862998
- [Derived] Di Gioia CC, Artusi N, Xotta G, Bonsano M, Sisto UG, Tecchiolli M, Orso D, Cominotto F, Amore G, Meduri S, Copetti R. Lung ultrasound in ruling out COVID-19 pneumonia in the ED: a multicentre prospective sensitivity study. Emerg Med J. 2022 Mar;39(3):199-205. doi: 10.1136/emermed-2020-210973. Epub 2021 Dec 22. PMID 34937709